CLINICAL TRIAL: NCT06979401
Title: Effects of Foot Sensory Training on Plantar Sensation, Functional Performance, Balance, Gait and Kinesiophobia in Type 2 Diabetic Individuals With Neuropathy
Brief Title: Effect of Sensory Training on Functional Performance, Balance, Gait in Type 2 Diabetic Individuals With Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aylin DEMİR (Other)
Responsible Party: Sponsor-Investigator, Aylin DEMİR, RESEARCH ASSISTANT, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/7046
Record Dates: First submitted 2025-05-10; First posted 2025-05-19 (Actual); Last update posted 2025-05-19 (Actual); Status verified 2025-05

CONDITIONS: Diabetes; Type 2 Diabetes; Diabetic Peripheral Neuropathy; Kinesiophobia; Balance; Functional Performance; Gait Analysis; Plantar Sensation
Keywords: balance; Plantar Sensation; type 2 diabetes; gait; kinesiophobia; functional performance; diabetic peripheral neurophaty
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Kinesiophobia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): After obtaining informed consent to participate in the study, all participants will be evaluated by an experienced physiotherapist before group allocation. All participants will receive diabetic foot training. Then, the intervention group and the control group will be formed by a sequential random method. Foot sensory training will be applied to the intervention group and no intervention will be made to the control group. However, after the study is completed, sensory training will be provided to the participants in the control group who wish to do so. Foot sensory training will be performed by the researcher physiotherapist. Foot sensory training sessions will be planned for 6 weeks, 3 days a week. An initial assessment will be made before the sessions begin and a final assessment will be made after the 6-week foot sensory training program.
  Interventions: Other: Exercise
- Control (No Intervention): Individuals who agree to participate in the study and meet the inclusion criteria will be asked for written consent with a consent form. The researcher will meet with the participants one-on-one and provide information about the purpose of the study. The pre-test data of the study will be collected by an experienced physiotherapist before group allocation. All participants will receive diabetic foot training. Then, the intervention group and the control group will be formed with a sequential random method. Individuals in the control group will not receive any intervention and will continue their standard drug treatments for diabetes. Post-test data will be collected after the 6-week sensory training given to the intervention group. They will only complete the pre-test and post-test and will not participate in sensory training. Their data will be used for comparison purposes to evaluate the effectiveness of the intervention.

INTERVENTIONS:
Other: Exercise — After obtaining informed consent to participate in the study, all participants will be evaluated by an experienced physiotherapist before group allocation. All participants will receive diabetic foot training. Then, the experimental group and the control group will be formed by a sequential random method. Foot sensory training will be applied to the experimental group and no intervention will be made to the control group. However, after the study is completed, sensory training will be provided to the participants in the control group who wish to do so. Foot sensory training will be performed by the researcher physiotherapist. Foot sensory training sessions will be planned for 6 weeks, 3 days a week. An initial assessment will be made before the sessions begin and a final assessment will be made after the 6-week foot sensory training program.
  Other Names: foot sensory training
  Arms: intervention

SUMMARY:
Diabetic peripheral neuropathy (DPN) is a common complication of type 1 and type 2 diabetes. DPN is characterized by significant axonal degeneration and segmental demyelination affecting sensory and motor nerves. The effect of foot sole sensation on gait and balance parameters has been reported in various studies in the literature, however, no study has been found examining the effect of foot sensory training on plantar sensation, functional performance, balance, gait and kinesiophobia in type 2 diabetic individuals with neuropathy. In order to contribute to the literature, 40 type 2 diabetic individuals with neuropathy who applied to the Turgut Ozal Medical Center Endocrinology and Metabolic Diseases Polyclinic will be included in this randomized controlled study. After diabetic foot training is given to all participants, an experimental (20) and a control (20) group will be formed with a sequential random method. Foot sensory training will be given to the experimental group, while no intervention will be made to the control group, and sensory training will be given to the participants who wish after the study is completed. All participants will be evaluated for subscapular sense, functional performance, balance, walking and kinesiophobia at the beginning and end of the training. Subscapular sense will be evaluated with light touch, two-point discrimination and vibration tests. Functional performance evaluation will be made with timed up and go test and timed stair ascent-descend test. Kinesiophobia will be analyzed with Tampa Kinesiophobia Scale, Balance; One-Legged Stand Test and Y balance tests and walking will be analyzed with Kinect V2 camera based software. Physical activity levels will be evaluated with International Physical Activity Questionnaire-Short Form. The data taken into the research will be analyzed with SPSS (Statistical Program in Social Sciences) program. The values belonging to the data will be expressed with percentage, mean and standard deviation, and the significance level (p) will be taken as 0.05 for comparison tests.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a chronic metabolic disease that develops as a result of insufficiency of insulin itself or its action. Diabetic peripheral neuropathy (DPN), a common complication of type 2 diabetes, results from metabolic and microvascular changes as a consequence of prolonged hyperglycemia and metabolic derangements.

Diabetic peripheral neuropathy is associated with damage to small unmyelinated and myelinated nerve fibers, resulting in impaired sensations of touch, pain and temperature. Damage to large myelinated nerve fibers results in decreased sensation of vibration and proprioception. Sole sensation is an important parameter for posture and gait control. When the afferent inputs of the foot are not properly transmitted to the central nervous system, a lack of balance develops reciprocally.

Functional performance refers to some activities and behaviors in daily life that individuals can perform up to a certain level. In individuals with diabetes mellitus with neuropathy, it is reported that there are decreases in functional performance as well as strength losses and decreases in joint mobility, especially in the dorsal and plantar foot muscles.

Involving both sensory and motor fibers, DPN causes balance and gait disturbances and neuropathic pain. As a result of altered gait biomechanics and balance disorders, individuals with diabetes have an increased risk of falling, perception of imbalance and fear of falling. This leads to physical inactivity and loss of muscle strength. It leads to further impairment of gait and balance biomechanics.

Kinesiophobia is the patient's fear of physical movement as well as negative cognitive and emotional response to anticipated or actual pain. It is expressed as a condition describing actions resulting from a feeling of vulnerability to re-injury. Impaired balance and fear of falling initiate kinesiophobia in people. As a result, restriction in physical activities increases. The number of studies examining kinesiophobia in individuals with diabetes is very limited. In one study, it was stated that individuals with diabetic neuropathy had an increase in kinesiophobia in balance disorders.

When the studies conducted with type 2 diabetic individuals with neuropathy were examined in the literature, no study providing foot sensory training was found. In this study, we aimed to investigate the effect of foot sensory training on underfoot sensation, functional performance, balance, gait and kinesiophobia in type 2 diabetic individuals with neuropathy. This study will provide data and contribution to fill this gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being 35-65 years old
* Being diagnosed with type 2 diabetes
* Having achieved glycemic control
* Having given less than 8 correct answers in the Semmes-Weinstein Monofilament test performed with a 5.07 monofilament
* Getting a Neuropathy Disability Score of 3 and above
* Being willing to participate in the study
* Being literate

Exclusion Criteria:

* Having a neurological or orthopedic comorbidity
* Having a respiratory disease such as uncontrolled COPD or asthma
* Having active lower extremity ulceration
* Using medications known to affect the postural control system such as benzodiazepines
* Having nephropathy, retinopathy and diabetic arthritis at a level that may affect mobility in addition to neuropathy
* Using a walking aid
* Body Mass Index >30
* Having communication problems
* Not participating in at least 3 consecutive exercise sessions
* Not participating in more than 30% of each session

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale | 6 week
  Tampa Kinesiophobia Scale is a Likert-type scale consisting of 17 questions. Turkish validity and reliability of the scale has been performed. It is used to determine the level of kinesiophobia of individuals.
Evaluation of Light touch sense | 6 week
  Light touch sensation will be evaluated using Semmes-Weinstein Monofilaments with reference to the metatarsal head, 5th metatarsal head and heel midpoint. The monofilament will be held for 1-1.5 seconds at each reference point and the patient will be asked to say "yes" when they feel the filament. 3 measurements will be taken from each point and 10 seconds will be allowed between measurements. The value of the filament felt by the patient will be recorded as a score.
Timed Up and Go Test | 6 week
  The timed get up and go test was developed to assess functional mobility parameters such as walking speed, postural control and balance. This test involves standing up from a normal-sized chair without arms, walking three meters, then returning and sitting back down on the chair. During the test, the individual will be asked to take a trial walk and then carefully perform the test three times. The average of these three tests will be taken as the basis. Walking speed will be recorded in seconds. The time will be started when the individual stands up from the chair. It will be stopped and recorded when the individual sits back in the chair.
Single Leg StanceTest | 6 week
  The Single Leg StanceTest will be used to assess static balance. For this test, participants will be asked to stand without falling for 30 s with the non-evaluated side knee in 90° flexion. The stopwatch will be started as soon as the foot leaves the ground. Each fall to maintain balance will be recorded as a score. The test will be repeated 3 times for the right and left lower extremities and averaged.
Gait Analysis | 6 week
  The gait analysis of the participants will be evaluated with a Kinect V2 camera-based software. This software is developed in MATLAB environment and identifies joint positions by processing depth images. In the developed software, the joint position is first determined for a pixel in the depth images and the accuracy level is calculated for each pixel. A validation study of the gait analysis of the Kinect camera system was conducted by Baldewijns et al.
Evaluation of vibration sense | 6 week
  The sense of vibration will be evaluated using a 128-Hz frequency diapason. Measurements will be made with the patient in the supine position with eyes closed, with reference to the 1st metatarsal head and medial malleolus. Each measurement point will be repeated three times and the average will be recorded in seconds.
Evaluation of Two-point discrimination sense | 6 week
  Two-point discrimination will be assessed using an esthesiometer. In the study, trans-metatarsal, heel midpoint and midfoot midpoint will be taken as reference. The esthesiometer will be touched sequentially to the reference points on the sole of the participant's foot. Measurement will start from the maximum distance and continue by decreasing the range. The distance at which the patient perceives one point instead of two points at the specified reference points will be recorded in millimeters.
Stair Climb Test | 6 week
  The stair climb test was developed to assess functional mobility content such as strength, speed and maneuverability. The test consists of the participant climbing the steps of the staircase and descending back to the starting point from the 10th step. They are free to hold on the edge of the ladder. At the beginning of the test, the participants will be asked to climb the ladder with a total of 10 steps and without waiting, turn back, descend the ladder and return to the starting point. During the test, the individual will be asked to perform a trial test. They will then be asked to repeat the test three times. These three tests will be averaged. Starting with the go command, the time in seconds will be recorded until both feet land on the floor on the return.
Y Balance test | 6 week
  The Y Balance Test will be used for the assessment of dynamic balance. After the individual is placed in the center of the Y-shaped apparatus with hands on the waist, they will be asked to reach in the anterior, posteromedial and posterolateral directions with the other leg with one leg fixed. While extending the moving foot along the desired vector throughout the measurement, they will be asked to touch the farthest point they can reach without losing their balance in a one-leg stance and the distance of this point to the center will be measured. Reaching will be asked 3 times in each direction and then the average of the reaching distances will be taken and recorded in centimeters. The test will be applied to both extremities.

CONTACTS AND LOCATIONS:
Locations (1):
- İnonu University, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No